CLINICAL TRIAL: NCT03025139
Title: Improving Outcomes for Younger Breast Cancer Survivors: A Phase III Randomized Trial Targeting Behavioral Symptoms in Younger Breast Cancer Survivors
Brief Title: Mindfulness Meditation or Survivorship Education in Improving Behavioral Symptoms in Younger Stage 0-III Breast Cancer Survivors (Pathways to Wellness)
Acronym: PTW
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 16-000817; NCI-2016-01396 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); R01CA200977 (NIH)
Record Dates: First submitted 2017-01-17; First posted 2017-01-19 (Estimated); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Cancer Survivor; Early-Stage Breast Carcinoma; Stage 0 Breast Cancer; Stage IA Breast Cancer; Stage IB Breast Cancer; Stage IIA Breast Cancer; Stage IIB Breast Cancer; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer
Keywords: breast cancer; younger women; education; mindfulness meditation; depression; cancer survivor
MeSH Terms: conditions — Breast Neoplasms; Breast Carcinoma In Situ; Depression | interventions — Early Intervention, Educational; Educational Status; Methods; Meditation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm A (MAPs) (Active Comparator): Patients attend a mindfulness meditation class over 2 hours once weekly for 6 weeks. Patients then attend in person booster sessions that include guided meditation, questions, and discussion of how to maintain a mindfulness practice over 1 hour once monthly for 2 months.
  Interventions: Other: Laboratory Biomarker Analysis; Procedure: Meditation Therapy; Other: Questionnaire Administration
- Arm B (SE) (Active Comparator): Patients attend a survivorship education class over 2 hours once weekly for 6 weeks. Patients also receive monthly electronic newsletters with tailored information about topics of interest to younger survivors, including cancer-related events in the community and tips about following through on recommendations for healthy living.
  Interventions: Other: Educational Intervention; Other: Laboratory Biomarker Analysis; Other: Questionnaire Administration
- Arm C (USUAL CARE/DELAYED TREATMENT CONTROL GROUP) (Active Comparator): Patients receive usual care for 9 months. Patients are then offered a choice of participating in Arm A or Arm B.
  Interventions: Other: Educational Intervention; Other: Laboratory Biomarker Analysis; Procedure: Meditation Therapy; Other: Questionnaire Administration

INTERVENTIONS:
Other: Educational Intervention — Attend survivorship education
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
  Arms: Arm B (SE); Arm C (USUAL CARE/DELAYED TREATMENT CONTROL GROUP)
Other: Laboratory Biomarker Analysis — Correlative studies
Procedure: Meditation Therapy — Attend mindfulness meditation
  Other Names: Meditation
  Arms: Arm A (MAPs); Arm C (USUAL CARE/DELAYED TREATMENT CONTROL GROUP)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This randomized phase III trial studies how well mindfulness meditation or survivorship education work in improving behavioral symptoms in younger stage 0-III breast cancer survivors. Behavioral interventions, such as mindfulness meditation, use techniques to help patients change the way they react to environmental triggers that may cause a negative reaction. Survivorship education after treatment may reduce stress and improve the well-being and quality of life of patients with breast cancer. Mindfulness meditation or survivorship education may help improve the health behaviors of younger breast cancer survivors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the efficacy of two different types of group interventions (mindfulness and survivorship education), specifically tailored to the needs of younger female breast cancer survivors, in reducing depressive symptoms, compared to a usual care control group.

SECONDARY OBJECTIVES:

I. To compare the efficacy of the two interventions relative to a usual care control group on fatigue, sleep disturbance, and vasomotor symptoms.

II. To examine the efficacy of the two interventions relative to a usual care control group on circulating and genomic markers of inflammation.

III. To explore potential moderators and mediators of intervention efficacy in the two intervention groups.

OUTLINE: Patients are randomized to 1 of 3 arms.

ARM A (MINDFULNESS AWARENESS PRACTICES [MAPs]): Patients attend a mindfulness meditation class over 2 hours once weekly for 6 weeks. Patients then attend in person booster sessions that include guided meditation, questions, and discussion of how to maintain a mindfulness practice over 1 hour once monthly for 3 months.

ARM B (SURVIVORSHIP EDUCATION INTERVENTION [SE]): Patients attend a survivorship education class over 2 hours once weekly for 6 weeks. Patients also receive monthly electronic newsletters with tailored information about topics of interest to younger survivors, including cancer-related events in the community and tips about following through on recommendations for healthy living.

ARM C (USUAL CARE/DELAYED TREATMENT CONTROL GROUP): Patients receive usual care for 9 months. Patients are then offered a choice of participating in Arm A or Arm B.

After completion of study, patients are followed up at 3 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed with early stage, resectable breast cancer (Stage 0, I, II, or III) prior to age 50, and are within 5 years of diagnosis
* Have completed all surgery, radiation, and/or chemotherapy treatments at least 6 months previously; may still be receiving trastuzumab or endocrine adjuvant therapy
* Ability to complete evaluation surveys in English
* Have evidence of at least mild clinical depression on a standardized screening questionnaire

Exclusion Criteria:

* Has a breast cancer recurrence, metastasis, or another interval cancer diagnosis following the breast cancer (excluding non-melanoma skin cancer)
* Unable to commit to intervention schedule (6 weekly group meetings)
* Actively practicing mindfulness meditation
* Has another serious or chronic medical or psychiatric condition that contributes to substantial physical or emotional disability that would detract from participating in either of the intervention programs or from the measurement of intervention outcomes

Max Age: 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 96 (Actual)
Dates: Start 2017-02-20 (Actual); Primary Completion 2023-02-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Change in depressive symptoms measured by Center for Epidemiologic Studies Depression Scale score | 2 weeks post-intervention to 6 months
  The data will be analyzed using linear mixed effects models, with fixed effects for time and condition and random effects for individuals. Differences between conditions in change over time will be examined by testing condition-by-time interaction terms. All tests will be two-sided. The Hochberg procedure will be applied to the two p-values for each intervention to control the familywise error rate at 0.05.

SECONDARY OUTCOMES:
Change in fatigue assessed by Fatigue Symptom Inventory | 2 weeks post-intervention to 6 months
  Will be tested using the mixed modeling approach, and p-values reported both with and without multiplicity adjustment. All tests will be two-sided.
Change in hot flashes measured by the vasomotor symptom severity subscale of the BCPT symptom scales questionnaire. | 2 weeks post-intervention to 6 months
  Will be tested using the mixed modeling approach, and p-values reported both with and without multiplicity adjustment. All tests will be two-sided.
Change in inflammatory biomarkers will focus on laboratory measurements of Interleukin-6 (IL-6) and high sensitivity C-Reactive Protein (hsCRP) | 2 weeks post-intervention to 6 months
  Will be tested using the mixed modeling approach, and p-values reported both with and without multiplicity adjustment. All tests will be two-sided.
Change in sleep disturbance assessed by Insomnia Severity Index | 2 weeks post-intervention to 6 months
  Will be tested using the mixed modeling approach, and p-values reported both with and without multiplicity adjustment. All tests will be two-sided.
Mediators of intervention efficacy assessed by questionnaire | Up to 6 months
  Mediators assessed will include self-efficacy, mindfulness, self-kindness, and rumination.
Moderators of intervention efficacy assessed by questionnaire | Up to 6 months
  Moderators will include preparedness for survivorship, intervention preference, and childhood adversity. Will be assessed using condition-by-moderator interaction terms in mixed models.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Ganz, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (3):
- United States (3):
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts

REFERENCES:
- [Derived] Korecki JRT, Ganz PA, Partridge AH, Wolff AC, Petersen L, Crespi CM, Bower JE. Mediators of a Mindfulness-Based Intervention for Younger Breast Cancer Survivors: Effects on Depressive Symptoms. Psychosom Med. 2024 Oct 1;86(8):700-709. doi: 10.1097/PSY.0000000000001340. Epub 2024 Aug 10. PMID 39132946
- [Derived] Tyrus Korecki JR, Ganz PA, Partridge AH, Wolff AC, Petersen L, Crespi CM, Bower JE. Moderators of Intervention Efficacy in the Pathways to Wellness Trial of Survivorship Education and Mindfulness Meditation for Younger Breast Cancer Survivors. JCO Oncol Pract. 2024 Oct;20(10):1410-1419. doi: 10.1200/OP.23.00617. Epub 2024 Jun 25. PMID 38917400
- [Derived] Bower JE, Partridge AH, Wolff AC, Cole SW, Irwin MR, Thorner ED, Joffe H, Petersen L, Crespi CM, Ganz PA. Improving biobehavioral health in younger breast cancer survivors: Pathways to Wellness trial secondary outcomes. J Natl Cancer Inst. 2023 Jan 10;115(1):83-92. doi: 10.1093/jnci/djac180. PMID 36130057
- [Derived] Bower JE, Partridge AH, Wolff AC, Thorner ED, Irwin MR, Joffe H, Petersen L, Crespi CM, Ganz PA. Targeting Depressive Symptoms in Younger Breast Cancer Survivors: The Pathways to Wellness Randomized Controlled Trial of Mindfulness Meditation and Survivorship Education. J Clin Oncol. 2021 Nov 1;39(31):3473-3484. doi: 10.1200/JCO.21.00279. Epub 2021 Aug 18. PMID 34406839

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-22): https://cdn.clinicaltrials.gov/large-docs/39/NCT03025139/Prot_SAP_000.pdf